CLINICAL TRIAL: NCT05196880
Title: A Prospective, Single-blind, Clinical Evaluation of the MolecuLight DX in Combination With Biofilm Based Wound Care for the Identification of Biofilm Containing Wounds
Brief Title: Biofilm Correlation and Validation
Status: Completed | Type: Observational
Sponsor: MolecuLight Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-002
Record Dates: First submitted 2021-12-14; First posted 2022-01-19 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- ARM 1: Patients with negative clinical suspicion of Biofilm containing wounds(CSB-).
  Interventions: Device: MolecuLight DX Imaging Device
- ARM 2: Patients with positive clinical suspicion of Biofilm containing wounds(CSB+)
  Interventions: Device: MolecuLight DX Imaging Device

INTERVENTIONS:
Device: MolecuLight DX Imaging Device — The MolecuLight DX Imaging Device is a fluorescence imaging device intended to acquire images from wounds. This will not alter the participant's standard of care treatment.

SUMMARY:
This is a prospective, single-blind, controlled trial. There are two arms and 20 patients with acute or chronic wounds with clinical suspicion of biofilm (CSB+/CSB-) are allocated in each arm. The primary objective is to evaluate the diagnostic accuracy of MolecuLight fluorescence in identifying biofilm as validated by gold standard SEM imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with acute or chronic wounds
2. 18 years or older
3. Willing to consent

Exclusion Criteria:

1. Treatment with an investigational drug within 1 month of enrolment
2. Any contra-indication to regular wound care
3. Inability or unwillingness to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects presenting with acute or chronic wounds
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of fluorescence signature to predict presence or absence of wound biofilm measured by moderate/ heavy bacterial load | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Mayer Institute, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided